CLINICAL TRIAL: NCT00213655
Title: Clinical Evaluation of Maintenance BCG Immunotherapy in Superficial Bladder Tumors
Brief Title: URO-BCG-4 : Bladder Tumors Immunotherapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2003/081/HP
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Daily instillation of BCG for 3 weeks then every 6 months: Effect of daily instillation of BCG (27 mg) for 3 weeks then one instillation of BCG (27 mg) every 6 months for 36 months on bladder tumor recurrence
  Interventions: Biological: bladder tumor recurrence
- Daily instillation of BCG for 2 weeks then every 3 months: Effect of daily instillation of BCG (27 mg) for 2 weeks then one instillation of BCG (27 mg) every 3 months for 36 months on bladder tumor recurrence
  Interventions: Biological: bladder tumor recurrence

INTERVENTIONS:
Biological: bladder tumor recurrence — bladder tumor recurrence assessed by clinical and biological exams

SUMMARY:
Evaluation of maintenance BCG immunotherapy (dose 27 mg) in superficial bladder tumors. Two randomized arms (every 3 or 6 months) will be studied for a population of 300 patients.

DETAILED DESCRIPTION:
BCG maintenance immunotherapy 1/3 dose : 27 mg two randomized arms : 3 or 6 months for 36 months clinical side effects according to OMS score efficacy regarding recurrence : cytology and cystoscopy PSA, leucocyturia and N-ramp gene evaluation

ELIGIBILITY:
Inclusion Criteria:

* Ta and T1 bladder tumors

Exclusion Criteria:

* BCG contra-indications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bladder Cancer
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2004-06; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Tumoral response | Month 36
  Tumoral response assessed at M36

SECONDARY OUTCOMES:
Tumoral response | Month 24
  Tumoral response assessed at M24

CONTACTS AND LOCATIONS:
Overall Officials: Christian PFISTER, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Charles Nicolle, University Hospital, Rouen, France